CLINICAL TRIAL: NCT06191432
Title: Tolerability of an Ancient Grain in Patients With Non-Celiac Wheat Sensitivity. A Clinical Study and a Search for Diagnostic Biomarkers.
Brief Title: Tolerability of an Ancient Grain in Patients With Non-Celiac Wheat Sensitivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Associate Professor, University of Palermo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: ACPM33
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Non-celiac Gluten Sensitivity
Keywords: Irritable Bowel Syndrome; Non-celiac wheat sensitivity; Triticum monococcum; Ancient grains
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, cross-over, single center clinical trials.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be assigned by a computerized algorithm to start the challenge with the sachets containing triticum monococcum or triticum aestivum. At the end of the first challenge and after an adequate wash-out period, the patients will undergo crossover with the other type of wheat sachets.
  The sachets, called A or B, will be completely indistinguishable from each other both in terms of their organoleptic characteristics and the quantity of content (80g of flour) and in terms of their packaging. The company that will supply the flours will be the custodian of the randomization code, and the key will be provided to the experimenters only at the end of all the challenges.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NCWS Packets A-B (Experimental): NCWS patients will undergo a Double-Blind Wheat Challenge DBWC with an ancient diploid wheat (TM) or a modern hexaploid wheat (TA). This DBWC will be performed with flour packets coded A or B, each containing respectively one of the wheat varieties. Packets A or B will be given for 1 week and then, after 1 week of washout (or until patients report complete well-being), the patients will receive the other packets for another 1 week (cross-over design).
  Interventions: Dietary Supplement: Administration of Triticum Monococcum flour; Dietary Supplement: Administration of Triticum Aestivum flour
- NCWS Packets B-A (Experimental): NCWS patients will undergo a Double-Blind Wheat Challenge DBWC with an ancient diploid wheat (TM) or a modern hexaploid wheat (TA). This DBWC will be performed with flour packets coded A or B, each containing respectively one of the wheat varieties. Packets A or B will be given for 1 week and then, after 1 week of washout (or until patients report complete well-being), the patients will receive the other packets for another 1 week (cross-over design).
  Interventions: Dietary Supplement: Administration of Triticum Monococcum flour; Dietary Supplement: Administration of Triticum Aestivum flour

INTERVENTIONS:
Dietary Supplement: Administration of Triticum Monococcum flour — Patients will be administered a daily dose of 80g of flour of Triticum Monococcum (equivalent to 10g of gluten), which will be dissolved and cooked by the patients themselves. During the challenge, the severity of the symptoms will be recorded using a 10-points visual analog scale (VAS). The challenges will be stopped when clinical reactions will occur for at least 2 consecutive days (increase >3 in VAS) for either GI or extraintestinal symptoms.
  Challenges will be considered positive if symptoms, which had been initially present, reappear after their disappearance on elimination diet, and if the GI and/or extraintestinal symptom's scores will be >30% compared to any eventual increase determined during the administration of the other wheat variety.
Dietary Supplement: Administration of Triticum Aestivum flour — Patients will be administered a daily dose of 80g of flour of Triticum Aestivum (equivalent to 10g of gluten), which will be dissolved and cooked by the patients themselves. During the challenge, the severity of the symptoms will be recorded using a 10-points visual analog scale (VAS). The challenges will be stopped when clinical reactions will occur for at least 2 consecutive days (increase >3 in VAS) for either GI or extraintestinal symptoms.
  Challenges will be considered positive if symptoms, which had been initially present, reappear after their disappearance on elimination diet, and if the GI and/or extraintestinal symptom's scores will be >30% compared to any eventual increase determined during the administration of the other wheat variety.

SUMMARY:
Patients suffering from wheat-related troubles, in absence of celiac disease or wheat allergy diagnosis, can suffer from non-celiac wheat sensitivity (NCWS). This is characterized by both gastrointestinal (GI) and extra-intestinal symptoms, which improve with the elimination of wheat intake. To date no definitive explanation of pathogenetic mechanisms of NCWS has been proved, and, similarly, no specific non-invasive diagnostic biomarker has been recognized. A real need of strict adherence to wheat-free diet (WFD) in NCWS has never been demonstrated. In this context, research is actively trying to find wheat varieties with absent or low immune-reactivity to be used for the treatment of NCWS patients. Preliminary evidence supports the assumption that diploid wheat species, as Triticum monococcum (TM), compared to common ones (Triticum aestivum (TA), could possess a lower immunogenic potential in NCWS patients. The first objective of our project is to verify whether the use of a diploid wheat (TM), with a lower concentrations and bioactivity of Amylase-Trypsin-Inhibitors (ATIs) and with gliadin proteins with a better digestibility, compared to a hexaploid one (TA) could improve both symptoms and quality of life (QoL) of NCWS subjects. The second objective is the identification of non-invasive serological biomarkers for NCWS diagnosis. The third objective is to identify T cell lymphocytes able to recognize cognate peptides from wheat proteins to better classify and monitor patients affected by NCWS. To achieve these results we planned a prospective, double-blind clinical trial with crossover, in which patients already diagnosed with NCWS (according to international criteria and with a double-blind placebo-controlled wheat challenge), following a strict WFD, will be exposed in double-blind to both TM and TA. All the patients will be evaluated clinically at the different timepoints with validated scales to assess tolerability of TM. Moreover, their intestinal permeability, immunological activation and gut microbiota patterns will be studied by both in vitro and in vivo techniques. Finally, a randomly chosen subset of patients will be studied through single cell transcriptome and T-cell receptor (TCR) sequencing on rectoscopy biopsy specimens to identify, T cell lymphocytes able to recognize cognate peptides from wheat proteins.

DETAILED DESCRIPTION:
State of the art The association between wheat intake and "wheat-related disorders" (WRDs) has been known for a long time, including pathologies as celiac disease (CD) and wheat allergy (WA). Recently a new non-allergic and non-autoimmune condition has been identified: non-celiac gluten sensitivity (NCGS). This is characterized by both gastrointestinal (GI) symptoms, very similar to those of irritable bowel syndrome (IBS) (eg. abdominal pain, diarrhea, etc.), and extra-intestinal ones (eg. arthromyalgias, anemia, etc.), which improve on a wheat-free diet (WFD).

NCGS prevalence rates range from 0.6% to 13% in the general population, and given the lack of a biomarker, its diagnosis is based on: 1) exclusion of CD and WA; 2) symptom's regression on a WFD; 3) recurrence of symptoms on a double-blind placebo-controlled challenge (DBPCC) with wheat.

Physicians recognize a significant overlap between NCGS and IBS and it is known that IBS affects about 25% of the general population. So, if a percentage of IBS patients could have benefit from a WFD, this would have a paramount impact on its social health costs, being estimated that its indirect costs (eg. loss of work and reduced productivity) are up to $20 billion/years in the US, with an annual cost of $9933 per patient. Furthermore, many patients with IBS-like or upper gastro-esophageal functional-like manifestations self-report a relationship between symptoms onset and wheat ingestion (wheat-intolerance). Nevertheless, a clinical approach with a WFD for all IBS patients would be unmotivated and dangerous, determining also a great economic burden.

In most IBS patients, visceral hypersensitivity may contribute to GI symptoms. Immune activation, due to mucosal mast cells (MCs) in close vicinity to gut nerves, appears to play a role in IBS symptom's onset. A possible neuro-immune interaction in the duodenal submucosa of NCGS patients involving MCs has been described, in order to explain GI symptoms. Other findings in NCGS include an increased infiltration of eosinophils in GI tract, which might produce several inflammatory (ie. eosinophil cationic protein (ECP) and tryptase) and neuromodulatory substances (eg. substance P and VIP).

Several studies have investigated the performance of serum biomarkers panels in differentiating IBS from NCGS and healthy subjects. These included inflammatory cytokines, chemokines, neurotransmitters and antibodies associated with CD. Therefore, it is critically important to investigate the performance of serum biomarkers panels to differentiate "real NCGS" from other conditions.

Having not definitively established whether gluten or some other wheat's component is responsible for symptom's triggering, NCGS has been renamed as non-coeliac wheat sensitivity (NCWS), which would exclude other relevant cereals, such as barley and rye. Some components of wheat other than gluten proteins could be potentially deleterious for NCWS patients, which include fermentable short-chain carbohydrates (FODMAPs) and amylase trypsin inhibitors (ATIs); the latter, activating toll-like receptor 4 complex in monocytes, macrophages and dendritic cells of the intestinal mucosa, might induce innate immunity in both CD and healthy subjects. Finally, some authors have focused on the activation of innate and/or acquired immunity, or gut microbiota modifications.

Research is actively trying to find wheat varieties with absent or low immune reactivity to be used to treat patients with NCWS. Preliminary evidence showed that diploid wheat species, as Triticum monococcum (TM), compared to common ones (Triticum aestivum (TA) and Triticum durum), could possess a lower immunogenic potential in NCWS and IBS patients. It seems that modern wheats contain higher concentrations and bioactivity of ATIs compared with diploid ones, and that gliadin from TM retain a reduced number of immunogenic peptides for CD patients due to a high in vitro digestibility. We found that ATIs from TM are sufficiently different than those from TA, so to determine lack of immune toxicity in CD after proteolytic digestion. Moreover, some data showed that in IBS the consumption of ancient wheat can reduce symptoms and proinflammatory cytokines and improves intestinal dysbiosis. In this context, we have recently shown that NCWS patients who consume ancient grains may receive a late diagnosis due to the possible clinical benefit (tolerability) obtained with these grains.

All these data, however, must be considered preliminary and the pathogenetic mechanisms and the real clinical tolerability of the ancient wheats remain to be confirmed. Thus, it is very important to evaluate the hypothesis that specific ancient wheat varieties could be tolerated and safe for NCWS patients, trying to identify, at the same time, possible non-invasive biomarkers to diagnose and differentiate NCWS from IBS patients.

Hypotheses and objectives Our hypothesis is that a dietary therapeutic approach based on the use of a diploid wheat (TM), with a lower concentrations and bioactivity of ATIs and with gliadin proteins with a better digestibility, could improve symptoms and quality of life (QoL) of NCWS patients.

We planned to perform a Double-Blind Wheat Challenge (DBWC), with crossover of 2 wheat varieties (TM vs TA), in patient diagnosed with NCWS according to Salerno criteria (6), to assess the putative clinical tolerability of TM, and analyze the immunological, intestinal permeability and microbial differences, trying to identify both the pathogenetic mechanisms and potential diagnostic biomarkers of NCWS, helping in distinguishing NCWS from IBS patients.

If confirmed, a dietary regimen with TM would be a more suitable and a less expensive alternative to a WFD, and the identification of a biomarker for NCWS will reduce the number of medical visits and examinations, with substantial economic savings for the national health systems. Furthermore, the putative beneficial effect of a diet based on a regional ancient wheat variety will contribute to the regional agriculture and food economy.

The overarching objective of the study is to investigate in NCWS patients if a challenge with an ancient wheat (TM) compared to a modern one (TA), have a lower symptom's response, reflecting visceral hypersensitivity, immune activation and distinct microbial profiles, in order to guarantee these patients a consistent alternative to WFD and increase their QoL.

The second objective is the identification of non-invasive serological biomarkers for NCWS diagnosis.

The third objective is to identify, through single cell (sc) transcriptome and T-cell receptor (TCR) sequencing, T cell lymphocytes able to recognize cognate peptides from wheat proteins to better classify patients affected by NCWS, with a translational relevance for future tailored therapies.

The experimental plan is divided into 4 work packages (WPs). Within each WP, a series of tasks have been defined.

WP1: evaluation of clinical response to TM compared to TA in NCWS patients by a DBWC with crossover.

Task 1.1: evaluation of GI symptoms evoked by dietary exposition to TM and TA by a validated GI symptoms rating scale.

Task 1.2: evaluation of extraintestinal symptoms evoked by dietary exposition to TM and TA by an extraintestinal symptoms rating scale.

Task 1.3: evaluation of QoL modifications determined by dietary exposition to TM and TA by a QoL validated scale.

WP2: evaluation of intestinal permeability and damage biomarkers in NCWS patients under 3 dietary regimens: WFD, TM and TA challenge.

Task 2.1: in vivo evaluation of intestinal permeability by the Lactulose/Mannitol (La/Ma) ratio test.

Task 2.2: analysis of serological indexes of intestinal damage and permeability, by ELISA assays.

WP 3: Evaluation of immunological, inflammatory, and visceral hypersensitivity response in NCWS patients under 3 dietary regimens: WFD, TM and TA challenge.

Task 3.1: analysis of fecal and plasmatic biomarkers of visceral hypersensitivity by ELISA assays.

Task 3.2: analysis of the humoral immune response to gluten by ELISA assays Task 3.3: analysis of serological inflammatory biomarkers by simultaneous high sensitivity microsphere-based Luminex technology and ELISA assays.

Task 3.4: immunophenotyping of whole blood for quantification of immune cell (IC) subpopulations and their activation status, evaluation of gut homing biomarkers and identification of specific cell population involved in the systemic immune response to wheat.

Task 3.5: Identification, through single cell (sc) transcriptome and TCR sequencing, of T cell lymphocytes able to recognize cognate peptides from wheat proteins, in the rectal mucosa of NCWS subjects.

WP4: evaluation of gut microbiota in NCWS patients under 3 different dietary regimens: WFD, TM and TA challenge.

Task 4.1: in vitro amplification of bacterial genetic materials from fecal samples by polymerase chain reaction (PCR) methods and identification of gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* age >18 and <65 years;
* negativity of class A (IgA) and G (IgG) immunoglobulin (Ig) anti-deamidated gliadin (anti-DGP); negativity of IgA and IgG anti-tissue transglutaminase (anti-tTG) and anti-endomysial antibodies (EMA) ;
* absence of intestinal villous atrophy, documented in all patients carrying the DQ2 and/or DQ8 human leukocyte antigen haplotypes (therefore regardless of the negativity of celiac disease-specific serum antibodies);
* absence of wheat allergy (negative prick test and/or serum IgE measurement specific to wheat, gluten and gliadin).

Exclusion Criteria:

* age <18 and >65 years;
* self-exclusion of gluten/wheat from the diet and refusal to reintroduce it, for diagnostic purposes, before entering the study;
* pregnancy;
* alcohol and/or drugs abuse;
* Helicobacter pylori and other bacterial and/or parasitic infections;
* diagnosis of chronic inflammatory intestinal diseases and other organic pathologies affecting the digestive system (for example, serious liver diseases), nervous system diseases, major psychiatric disorders, immunological deficits and impairments that limit physical activity;
* cancer
* patients undergoing chemotherapy and/or radiotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of gastrointestinal symptoms evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  A modified version of Gastrointestinal Symptom Rating Scale (GSRS) will be administered to all the patients during each outpatient visit to assess gastrointestinal symptoms before the challenge (T0, wheat free diet) and after exposure to both Triticum Monococcum (TM) and Triticum Aestivum (TA).
  Difference will be considered relevant if GSRS will be recorded >30% compared to T0 and/or to any eventual increase determined during the administration of the other wheat variety.
Evaluation of extraintestinal symptoms evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  A extraintestinal symptoms rating scale, based on the symptoms most frequently observed in NCWS patients, will be administered to all the patients during each outpatient visit to assess gastrointestinal symptoms before the challenge (T0, wheat free diet) and after exposure to both Triticum Monococcum (TM) and Triticum Aestivum (TA).
  Difference will be considered relevant if extraintestinal symptoms rating scale will be recorded >30% compared to T0 and/or to any eventual increase determined during the administration of the other wheat variety.
Evaluation of quality of life modification evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  The Irritable Bowel Syndrome-Quality of Life (IBS-QoL) will be used to assess patient's QoL. It is an already validated condition-specific tool for IBS patients, which incorporates specific subdomains, such as food avoidance, bowel habits, and the effect on the social/sexual relationships.
  IBS-QoL will be administered to all the patients during each outpatient visit to assess gastrointestinal symptoms before the challenge (T0, wheat free diet) and after exposure to both Triticum Monococcum (TM) and Triticum Aestivum (TA).
  Difference will be considered relevant if IBS-QoL will be recorded >30% compared to T0 and/or to any eventual increase determined during the administration of the other wheat variety.

SECONDARY OUTCOMES:
In vivo evaluation of intestinal permeability modification evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  In vivo evaluation of intestinal permeability will be performed using the Lactulose/Mannitol (La/Ma) ratio test, which has already been validated for gluten-related disorders, and other GI diseases with diarrhea and malabsorption. The test is based on the oral administration (after 12 hours of fasting) of an aqueous isosmolar solution (270mOsm) of 2 non-absorbable sugars (5g lactulose and 2g mannitol), in 150ml of water. Not being metabolizable, the 2 sugars are filtered by the kidneys and found in the urine; a urine collection for 5 hours after the bolus contains everything that has been filtered, with a La/Ma ratio <0.035, which is considered the "normal" intestinal permeability index (values ≥0.035 will be considered as index of increased GI permeability).
  La/Ma ratio difference will be considered relevant for p<0.05 compared to T0 values and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of serological indexes of intestinal permeability evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: zonulin | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Zonulin dosage will be performed by commercial ELISA kits according to the manufacturer's instructions.
  Zonulin values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of serological indexes of intestinal permeability evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: occludin | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Occludin dosage will be performed by commercial ELISA kits according to the manufacturer's instructions.
  Occludin values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of serological indexes of intestinal permeability evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: claudin 1 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Claudin 1 dosage will be performed by commercial ELISA kits according to the manufacturer's instructions.
  Claudin 1 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of serological indexes of intestinal injury evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: intestinal fatty acid-binding protein | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  intestinal fatty acid-binding protein dosage will be performed by commercial ELISA kits according to the manufacturer's instructions.
  intestinal fatty acid-binding protein values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of serological indexes of intestinal injury evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: lipopolysaccharide | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  lipopolysaccharide dosage will be performed by commercial ELISA kits according to the manufacturer's instructions.
  lipopolysaccharide values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of serological indexes of intestinal injury evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: lipopolysaccharide binding-protein | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  lipopolysaccharide binding-protein dosage will be performed by commercial ELISA kits according to the manufacturer's instructions.
  lipopolysaccharide binding-protein values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of serological indexes of intestinal injury evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: F-actin immunoglobulin (Ig)A | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  F-actin immunoglobulin (Ig)A dosage will be performed by commercial ELISA kits according to the manufacturer's instructions.
  F-actin immunoglobulin (Ig)A values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of serological indexes of intestinal injury evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: F-actin immunoglobulin (Ig)G | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  F-actin immunoglobulin (Ig)G dosage will be performed by commercial ELISA kits according to the manufacturer's instructions.
  F-actin immunoglobulin (Ig)G values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of gut hypersensitivity indexes evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: eosinophil cationic protein | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Eosinophil cationic protein dosage will be performed on stool samples following already validated methodologies.
  Eosinophil cationic protein values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of gut hypersensitivity indexes evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: tryptase | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Tryptase dosage will be performed on stool samples following already validated methodologies.
  Tryptase values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of gut hypersensitivity indexes evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: substance P | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Substance P dosage will be performed on blood samples by commercial ELISA kits according to the manufacturer's instructions.
  Substance P values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of gut hypersensitivity indexes evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: somatostatin | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Somatostatin dosage will be performed on blood samples by commercial ELISA kits according to the manufacturer's instructions.
  Somatostatin values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of gut hypersensitivity indexes evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: serotonin | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Serotonin dosage will be performed on blood samples by commercial ELISA kits according to the manufacturer's instructions.
  Serotonin values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of gut hypersensitivity indexes evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: vasoactive intestinal peptide | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Vasoactive intestinal peptide dosage will be performed on blood samples by commercial ELISA kits according to the manufacturer's instructions.
  Vasoactive intestinal peptide values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the humoral immune response to gluten evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: anti-gliadin antibodies immunoglobulin A | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Humoral immune response to gluten will be evaluated by dosing plasmatic levels of anti-gliadin antibodies immunoglobulin A by commercial ELISA assays, following manufacturer's instructions.
  Anti-gliadin antibodies immunoglobulin A values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the humoral immune response to gluten evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: anti-gliadin antibodies immunoglobulin G | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Humoral immune response to gluten will be evaluated by dosing plasmatic levels of anti-gliadin antibodies immunoglobulin G by commercial ELISA assays, following manufacturer's instructions.
  Anti-gliadin antibodies immunoglobulin G values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: granulocyte colony-stimulating factor | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  Granulocyte colony-stimulating factor values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: granulocyte-macrophage colony-stimulating factor | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  Granulocyte-macrophage colony-stimulating factor values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interferon (IFN)-γ | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  Interferon (IFN)-γ values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-1β | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-1β values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-2 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-2 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-4 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-4 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-5 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-5 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-6 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-6 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-8 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-8 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-9 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-9 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-10 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-10 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-12 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-12 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-13 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-13 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-15 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-15 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-17 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-17 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-21 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-21 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-22 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-22 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: interleukin (IL)-33 | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  interleukin (IL)-33 values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of modification of the serological inflammatory biomarkers evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum: tumor necrosis factor (TNF)-α | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Expression of serological inflammatory biomarkers will be evaluated, on all the samples collected, by multiplexing simultaneous analysis with high sensitivity microsphere-based assays or ELISA.
  Tumor necrosis factor (TNF)-α values difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Analysis of immunophenotyping of whole blood for quantification of immune cell (IC) subpopulations modification and their activation status evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  Immunophenotyping will be performed by multi-color flow cytometry. Blood will be stained with fluorochrome conjugated antibodies specific for surface markers of cell population lineages and immune activation to allow the quantification of immune cell populations and their activation status Immune cell populations difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.
Identification of T cell lymphocytes able to recognize cognate peptides from wheat proteins | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  To identify T cells able to recognize cognate peptides from wheat proteins, CD45+ immune cells will be collected from rectal biopsy specimens obtained from 10 patients, at baseline and when they will report symptom's recurrence on double-blind wheat challenge. Rectal biopsies will be transferred in complete culture medium, minced into small pieces, followed by enzymatic digestion. Then CD45+ fraction will be sorted and used for subsequent -omic analyses. Immune cells obtained from the biopsies will undergo Single Cell characterization, aiming to investigate changes in the immune microenvironment, by CITE-seq and TCR-seq analyses. To gain insight into T Cell Receptor sequences able to recognize putative peptides originated from the main wheat proteins (gluten, etc.), we will develop a neural network/docking predictive model for TCR/epitope interaction. The final wheat peptides candidates will be then validated in vitro by using an Elispot assay.
Analysis of gut microbiota modification evoked by dietary exposition to Triticum Monococcum and Triticum Aestivum | Days 0 (before start of challenge), 7 (after intake of first kind of flour according randomization) and 21 (after intake of second kind of flour according randomization)
  in vitro identification of gut microbiota will be performed by amplification, analysis and quantification of gut microbiome on stools samples. After fecal collection, bacterial DNA will be extracted by cetyltrimethyl ammonium bromide, and 16S rDNA sequencing will be performed by polymerase chain reaction (PCR) methods, using universal primers. The resulting fragments will be then sequenced by pyrosequencing. Each reading will be compared with a database of known 16S rDNA sequences, using the BLAT program by phylogenetically assigning the most specific and reliable nodes. This method of assigning the obtained data leads to a "weighted" phylogenetic tree that characterizes well the bacterial content of the sample.
  Gut microbiota difference will be considered relevant for p<0.05 compared to values registered at T0 and/or to the values determined during the administration of the other wheat variety.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, MD, Study Chair — University of Palermo
Locations (1):
- University Hospital of Palermo, Palermo, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schuppan D, Pickert G, Ashfaq-Khan M, Zevallos V. Non-celiac wheat sensitivity: differential diagnosis, triggers and implications. Best Pract Res Clin Gastroenterol. 2015 Jun;29(3):469-76. doi: 10.1016/j.bpg.2015.04.002. Epub 2015 May 8. PMID 26060111
- [Result] Carroccio A, Giannone G, Mansueto P, Soresi M, La Blasca F, Fayer F, Iacobucci R, Porcasi R, Catalano T, Geraci G, Arini A, D'Alcamo A, Villanacci V, Florena AM. Duodenal and Rectal Mucosa Inflammation in Patients With Non-celiac Wheat Sensitivity. Clin Gastroenterol Hepatol. 2019 Mar;17(4):682-690.e3. doi: 10.1016/j.cgh.2018.08.043. Epub 2018 Aug 21. PMID 30138736
- [Result] Dieterich W, Schuppan D, Schink M, Schwappacher R, Wirtz S, Agaimy A, Neurath MF, Zopf Y. Influence of low FODMAP and gluten-free diets on disease activity and intestinal microbiota in patients with non-celiac gluten sensitivity. Clin Nutr. 2019 Apr;38(2):697-707. doi: 10.1016/j.clnu.2018.03.017. Epub 2018 Apr 4. PMID 29653862
- [Result] Rotondi Aufiero V, Fasano A, Mazzarella G. Non-Celiac Gluten Sensitivity: How Its Gut Immune Activation and Potential Dietary Management Differ from Celiac Disease. Mol Nutr Food Res. 2018 May;62(9):e1700854. doi: 10.1002/mnfr.201700854. Epub 2018 Apr 20. PMID 29578652
- [Result] Sofi F, Whittaker A, Gori AM, Cesari F, Surrenti E, Abbate R, Gensini GF, Benedettelli S, Casini A. Effect of Triticum turgidum subsp. turanicum wheat on irritable bowel syndrome: a double-blinded randomised dietary intervention trial. Br J Nutr. 2014 Jun 14;111(11):1992-9. doi: 10.1017/S000711451400018X. Epub 2014 Feb 13. PMID 24521561
- [Result] Seidita A, Mansueto P, Giuliano A, Chiavetta M, Mandreucci F, Soresi M, Pistone M, Compagnoni S, Castellucci D, Bisso G, Faraci F, Maestri S, Disclafani R, Sapone A, Fasano A, Carroccio A. Potential tolerability of ancient grains in non-celiac wheat sensitivity patients: A preliminary evaluation. Front Med (Lausanne). 2022 Sep 28;9:995019. doi: 10.3389/fmed.2022.995019. eCollection 2022. PMID 36250065